CLINICAL TRIAL: NCT00218231
Title: Transdermal Nicotine and Bupropion-SR in Schizophrenics (Study 2)
Brief Title: Effect of Bupropion on Smoking Behavior in Smokers With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jennifer W. Tidey, Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-14002-2; R01-14002-2; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia; Tobacco Use Disorder
Keywords: schizophrenia; tobacco dependence; nicotine
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 300 mg/day bupropion-sr
  Interventions: Drug: 300 mg/day bupropion-sr
- 2 (Placebo Comparator): 0 mg bupropion-sr
  Interventions: Drug: 0 mg/day bupropion-sr

INTERVENTIONS:
Drug: 300 mg/day bupropion-sr — 300 mg/day for 1 week
  Other Names: zyban, wellbutrin
  Arms: 1
Drug: 0 mg/day bupropion-sr — 0 mg/day bupropion-sr
  Other Names: placebo
  Arms: 2

SUMMARY:
Many individuals with schizophrenia smoke cigarettes but little is known about the factors that control smoking in people with schizophrenia. The purpose of this trial is to evaluate how bupropion, an antidepressant medication, affects smoking behaviors in individuals with schizophrenia who smoke.

DETAILED DESCRIPTION:
There is a high prevalence of cigarette smoking among people with schizophrenia and few smoking cessation interventions have been developed for these individuals. Bupropion is an antidepressant medication commonly used to treat smoking in smokers without psychiatric disorder. This study compares how smokers with schizophrenia and smokers without psychiatric illness respond to bupropion (0, 300 mg/day).

Participants will be randomly assigned to receive either bupropion or placebo. Study visits will occur after one-week treatment with placebo or bupropion. During study sessions, participants will come to the laboratory at 9 am and will remain abstinent in the laboratory for 5 hrs. Participants will then be assessed for craving and withdrawal symptoms after viewing and handling neutral cues and smoking cues. After that, participants will have a 90-min period to smoke, and smoking topography will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia or schizo-affective disorder
* Smokes between 20 and 50 cigarettes per day
* Moderate to high nicotine dependence score
* Interest in quitting smoking

Exclusion Criteria:

* Currently trying to quit smoking
* Seizure disorder or lowered seizure threshold due to anorexia, bulimia, head trauma, diabetes with insulin, or hypoglycemics
* Alcohol or drug use disorders
* Requires certain medications
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Smoking behavior | after 5 hrs abstinence

SECONDARY OUTCOMES:
Adverse events | ongoing
urge to smoke | after 5 hrs abstinence
nicotine withdrawal symptoms | after 5 hrs withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W. Tidey, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Providence VA Medical Center, RI, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961